CLINICAL TRIAL: NCT01286350
Title: FL3X: An Adaptive Intervention to Improve Outcomes for Youth With Type 1 Diabetes
Brief Title: FL3X Study: An Adaptive Intervention to Improve Outcomes for Youth With Type 1 Diabetes (FL3X)
Acronym: FL3X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Hospital Medical Center, Cincinnati (Other); University of Colorado, Denver (Other); University of Washington (Other); Nemours Children's Clinic (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2856 (UNC IRB); 1UC4DK101132-01 (NIH)
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: motivational interviewing; problem solving skills training; family communication; social support; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Participants randomized control will continue with usual clinical care.
- Intervention (Experimental): Participants randomized to intervention will receive the "FL3X Flexible Lifestyle Empowering Change" intervention. Adolescents will be paired with a health coach to help learn strategies for improving diabetes control
  Interventions: Behavioral: FL3X: Flexible Lifestyle Empowering Change

INTERVENTIONS:
Behavioral: FL3X: Flexible Lifestyle Empowering Change — The FL3X Adaptive Intervention is designed to increase adherence to T1D self-management including medical management (blood sugar testing and insulin dosing), diet, and physical activity. FL3X relies on MI, and problem-solving skills training (PSST) as the basis for the counseling strategy, and creates a coherent integration across three key components of 1) behavior family systems therapy focused on family communications and teamwork; 2) individualized diabetes education in response to knowledge gaps relevant to behavioral goal attainment; and 3) use of currently available communications technology to support behavioral goal attainment through participant-defined reminders and motivational boosters, and/or peer support.
  Other Names: FL3X
  Arms: Intervention

SUMMARY:
The purpose of this study is to see if a behavioral intervention for adolescents with type 1 diabetes will improve adherence to T1D self-management activities and improve diabetes outcomes. We expect the intervention to improve diabetes outcomes when compared to usual care.

DETAILED DESCRIPTION:
The FL3X Adaptive Intervention is designed to increase adherence to T1D self-management including medical management (blood sugar testing and insulin dosing), diet, and physical activity. FL3X relies on MI, and problem-solving skills training (PSST) as the basis for the counseling strategy, and creates a coherent integration across three key components of 1) behavior family systems therapy focused on family communications and teamwork; 2) individualized diabetes education in response to knowledge gaps relevant to behavioral goal attainment; and 3) use of currently available communications technology to support behavioral goal attainment through participant-defined reminders and motivational boosters, and/or peer support.

All FL3X intervention participants will receive "FL3X-Basic", which is the initial 3-month intervention that includes 4 sessions (40-60 min), supplemented with short additional contacts (via text, email, or web-based communication) as needed. Thereafter, applying principles of adaptive interventions, based on a decision rule using A1c values measured at defined intervals, participants are iteratively assigned to "FL3X-Check-in" or "FL3X-Regular", both of which continue with MI and PSST for the underlying counseling strategy. In FL3X-Check-in, participants who are doing well ("responders") will receive minimal ongoing support to reinforce successful strategies through brief monthly "touch-base" contacts. In FL3X-Regular, those who are "Regular-responders" will have a minimum of 3-4 in-person full-length sessions (40-60 min) over each 6-month interval, with additional brief contacts as needed (e.g., text, voice, or internet). FL3X participants randomized to the control group will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes with duration at least 12 months
* between ages 12-16 years at registration
* poor glycemic control (A1c 8.0-13.0%)
* parent/guardian willing to also participate
* not planning on moving in the following 18 months

Exclusion Criteria:

* pregnant (if female)
* diabetes type 2 or gestational
* Pre-existing systemic chronic disease (drug abuse, cancer, certain psychiatric conditions)

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 0, 3, 6, 12, 18, 24, 30 months
  HbA1c will be measured to determine impact on glucose control

SECONDARY OUTCOMES:
Motivation | 0, 3, 6, 12, 18, 24, 30 months
  Motivation related to diabetes care will be assessed
Problem solving skills | 0, 3, 6, 12, 18, 24, 30 months
  Assess use of problem solving skills relative to diabetes care
Hypoglycemia | 0, 6, 18 mo
  Monitoring low blood sugar from continuous glucose monitoring
Diabetes self-management behaviors | 0, 3, 6, 12, 18, 24, 30 months
  Assess use of diabetes self-management behaviors
Risk factors for diabetes complications | 0, 3, 6, 12, 18, 24, 30 months
  Assess variables related to diabetes complications
Health-related quality of life | 0, 3, 6, 12, 18, 24, 30 months
  Assess health-related quality of life

OTHER OUTCOMES:
Cost of intervention delivery | 0-30 months
  The study will evaluate cost to deliver intervention compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mayer-Davis, PhD, Principal Investigator — UNC-CH
Locations (2):
- United States (2):
  - University of Colorado Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Cristello Sarteau A, Crandell J, Seid M, Kichler JC, Maahs DM, Wang J, Mayer-Davis E. Characterization of youth goal setting in the self-management of type 1 diabetes and associations with HbA1c: The Flexible Lifestyle Empowering Change trial. Pediatr Diabetes. 2020 Nov;21(7):1343-1352. doi: 10.1111/pedi.13099. Epub 2020 Sep 1. PMID 32741045
- [Derived] Kahkoska AR, Lawson MT, Crandell J, Driscoll KA, Kichler JC, Seid M, Maahs DM, Kosorok MR, Mayer-Davis EJ. Assessment of a Precision Medicine Analysis of a Behavioral Counseling Strategy to Improve Adherence to Diabetes Self-management Among Youth: A Post Hoc Analysis of the FLEX Trial. JAMA Netw Open. 2019 May 3;2(5):e195137. doi: 10.1001/jamanetworkopen.2019.5137. PMID 31150087
- [Derived] Mayer-Davis EJ, Maahs DM, Seid M, Crandell J, Bishop FK, Driscoll KA, Hunter CM, Kichler JC, Standiford D, Thomas JM; FLEX Study Group. Efficacy of the Flexible Lifestyles Empowering Change intervention on metabolic and psychosocial outcomes in adolescents with type 1 diabetes (FLEX): a randomised controlled trial. Lancet Child Adolesc Health. 2018 Sep;2(9):635-646. doi: 10.1016/S2352-4642(18)30208-6. Epub 2018 Jul 30. PMID 30119757
- [Derived] Zhong VW, Crandell JL, Shay CM, Gordon-Larsen P, Cole SR, Juhaeri J, Kahkoska AR, Maahs DM, Seid M, Forlenza GP, Mayer-Davis EJ. Dietary intake and risk of non-severe hypoglycemia in adolescents with type 1 diabetes. J Diabetes Complications. 2017 Aug;31(8):1340-1347. doi: 10.1016/j.jdiacomp.2017.04.017. Epub 2017 Apr 20. PMID 28476567
- [Derived] Mayer-Davis EJ, Seid M, Crandell J, Dolan L, Lagarde WH, Letourneau L, Maahs DM, Marcovina S, Nachreiner J, Standiford D, Thomas J, Wysocki T. Flexible Lifestyles for Youth (FL3X) behavioural intervention for at-risk adolescents with Type 1 diabetes: a randomized pilot and feasibility trial. Diabet Med. 2015 Jun;32(6):829-33. doi: 10.1111/dme.12641. Epub 2014 Dec 30. PMID 25424501